CLINICAL TRIAL: NCT02238119
Title: A Randomised, Double-blind, Double-dummy, Crossover Efficacy and Safety Comparison of 6-week Treatment Periods of the Free Combination of Tiotropium Inhalation Powder Capsule (18 μg) + Formoterol Inhalation Powder Capsule (12 μg) QD, Tiotropium Inhalation Powder Capsule (18 μg) QD and Formoterol Inhalation Powder Capsule (12 μg) BID in Patients With COPD
Brief Title: Efficacy and Safety of Free Combination of Tiotropium + Formoterol Compared to Formoterol and Tiotropium in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1184.3
Record Dates: First submitted 2014-09-11; First posted 2014-09-12 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; Formoterol Fumarate

ARMS (3):
- tiotropium + formoterol (Experimental)
  Interventions: Drug: Tiotropium + formoterol combination
- tiotropium (Active Comparator)
  Interventions: Drug: Tiotropium
- formoterol (Active Comparator)
  Interventions: Drug: Formoterol

INTERVENTIONS:
Drug: Tiotropium + formoterol combination
  Arms: tiotropium + formoterol
Drug: Tiotropium
  Arms: tiotropium
Drug: Formoterol
  Arms: formoterol

SUMMARY:
Study to evaluate the lung function response to the free once-daily combination of tiotropium + formoterol compared to formoterol BID and tiotropium QD

ELIGIBILITY:
Inclusion Criteria:

1. All patients had to sign an informed consent consistent with International Conference on Harmonization Good Clinical Practice (ICH-GCP) guidelines prior to participation in the trial, which included medication washout and restrictions
2. All patients had to have a diagnosis of chronic obstructive pulmonary disease and had to meet the following spirometric criteria:

   * Patients had to have relatively stable moderate to severe airway obstruction with an FEV1 ≤ 60% of predicted normal and FEV1 ≤ 70% of FVC (Visits 1 and 2)
3. Male or female patients 40 years of age or older
4. Patients had to be current or ex-smokers with a smoking history of more than 10 pack-years (Patients who had never smoked cigarettes had to be excluded)
5. Patients had to be able to perform technically acceptable pulmonary function tests and had to be able to maintain records (Patient Daily Diary Record) during the study period as required in the protocol
6. Patients had to be able to inhale medication in a competent manner from the HandiHaler® device, the Blue Inhaler device and from a metered dose inhaler (MDI)

Exclusion Criteria:

1. Patients with significant diseases other than COPD had to be excluded. A significant disease was defined as a disease which in the opinion of the investigator may either put the patient at risk because of participation in the study or a disease which may influence the results of the study or the patient's ability to participate in the study
2. Patients with clinically relevant abnormal baseline haematology, blood chemistry, or urinalysis if the abnormality defined a disease listed as an exclusion criterion
3. All patients with an serum glutamate oxaloacetate transaminase (SGOT) > 80 IU/L, serum glutamate pyruvate transaminase (SGPT) > 80 IU/L, bilirubin > 17 μmol/L or creatinine > 110 μmol/L (males) / 95 μmol/L (females) had to be excluded regardless of clinical condition
4. Patients with a recent history (i.e., six months or less) of myocardial infarction
5. Patients with any cardiac arrhythmia requiring drug therapy or who had been hospitalised for heart failure within the past three years
6. Patients with a history of cancer within the last five years. Patients with treated basal cell carcinoma were allowed
7. Patients with known symptomatic prostatic hypertrophy or bladder neck obstruction.

   Patients with prostatic hypertrophy controlled by medication were allowed
8. Patients with known narrow-angle glaucoma
9. Patients with a history of asthma, allergic rhinitis or who had a total blood eosinophil count ≥600 mm3
10. Patients with a history of life-threatening pulmonary obstruction, or a history of cystic fibrosis or clinically evident bronchiectasis
11. Patients with known active tuberculosis
12. Patients with a history of and/or active significant alcohol or drug abuse. See exclusion criterion No. 1.
13. Patients who had undergone thoracotomy with pulmonary resection. Patients with a history of thoracotomy for other reasons had to be evaluated as per exclusion criterion No. 1
14. Patients who completed a pulmonary rehabilitation program in the six weeks prior to the Screening Visit (Visit 1)
15. Patients who regularly used daytime oxygen therapy
16. Patients who had taken an investigational drug within one month or six half lives (whichever is greater) prior to Screening Visit (Visit 1)
17. Patients who were treated with beta-blocker medications. Note: cardioselective beta blocker eye medications (e.g. Betoptic®) for treatment of non-narrow angle glaucoma were allowed
18. Patients who were treated with oral beta-adrenergics
19. Patients who were treated with cromolyn sodium or nedocromil sodium
20. Patients who were treated with antihistamines (H1 receptor antagonists), antileukotrienes or leukotriene receptor antagonists for asthma or excluded allergic conditions. See exclusion criterion No. 9
21. Patients using oral corticosteroid medication at unstable doses (i.e., less than six weeks on a stable dose) or at doses in excess of the equivalent of 10 mg of prednisone per day or 20 mg every other day
22. Patients with known hypersensitivity to anticholinergic drugs, beta-adrenergics, lactose or any other components of the inhalation capsule delivery systems
23. Pregnant or nursing women or women of childbearing potential not using a medically approved means of contraception for the previous 3 months (i.e. oral contraceptives, intrauterine devices, diaphragm or subdermal implants e.g., Norplant®)
24. Patients with previous participation (receipt of randomised treatment) in this study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2002-02; Primary Completion 2002-08 (Actual)

PRIMARY OUTCOMES:
Change in area under the curve from pre-dose to 12 hours of the forced expiratory volume in one second (FEV1 AUC0-12h) | after 6 weeks of each treatment
Change in FEV1 AUC0-24h | after 6 weeks of each treatment

SECONDARY OUTCOMES:
Change in FEV1 AUC12-24h | after 6 weeks of each treatment
Change in AUC of the forced vital capacity (FVC AUC0-12h) | after 6 weeks of each treatment
Change in FVC AUC0-24h | after 6 weeks of each treatment
Change in FVC AUC12-24h | after 6 weeks of each treatment
Change in peak FEV1 response | after 6 weeks of each treatment
Change in trough FEV1 response | after 6 weeks of each treatment
Change in peak FVC response | after 6 weeks of each treatment
Change in trough FVC response | after 6 weeks of each treatment
Individual FEV1measurements at each time point | up to 6 weeks
Individual FVCmeasurements at each time point | up to 6 weeks
Peak expiratory flow rate (PEFR) | weeks 4 to 6 of each treatment period
  measured twice daily
Number of inhalations of rescue salbutamol therapy used per day | weeks 4 to 6 of each treatment period
Assessment of daytime COPD symptom score rated on a 6-point rating scale | weeks 4 to 6 of each treatment period
Assessment of nighttime COPD symptom score rated on a 5-point rating scale | weeks 4 to 6 of each treatment period
Number of patients with adverse events | up to 23 weeks